CLINICAL TRIAL: NCT02729649
Title: ArmAssist Robotic Device for Arm Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Konstantinovic Ljubica, professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LK-3
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Hemiparesis
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ArmAssist therapy (Experimental): The group will be treated with ArmAssist robot therapy.
  Interventions: Device: ArmAssist robotic training; Other: Conventional therapy
- Conventional therapy (Active Comparator): The group will be treated with conventional therapy.
  Interventions: Other: Conventional therapy
- Extended Conventional therapy (Active Comparator): The group will be treated with extended conventional therapy.
  Interventions: Other: Conventional therapy; Other: Extended conventional therapy

INTERVENTIONS:
Device: ArmAssist robotic training
  Arms: ArmAssist therapy
Other: Conventional therapy
Other: Extended conventional therapy
  Arms: Extended Conventional therapy

SUMMARY:
ArmAssist is low cost simply robotic devise for arm training and assessment. It is suitable for extended home rehabilitation and prolonged hospital rehabilitation without therapist supervision. The device contains several games which are structured as exercise for disabled patients. The primary aim of this study is to correlate efficacy of the arm training with ArmAssist robot system to conventional care modified by duration and structure of exercise. The secondary aim of this study is to measure the correlation between standard clinical assessment scales and ArmAssist-based assessment metrics.

ELIGIBILITY:
Inclusion Criteria:

* unilateral paresis;
* ability to understand and follow simple instructions;
* minimum ability to perform active movements, even though trunk compensation, using the shoulder and/or the elbow joints.

Exclusion Criteria:

* bilateral impairment;
* severe sensory deficits in the paretic upper limb;
* cognitive impairment or behavioral dysfunction that would influence the ability to understand or perform the experiment;
* inability to provide informed consent;
* other current severe medical problems.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fugl Mayer motor score for upper extremity | 4 weeks

SECONDARY OUTCOMES:
Ashworth score | 4 weeks
Action research arm score | 4 weeks
Wolf motor function test | 4 weeks
Barthel index | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for rehabilitation dr Miroslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia

REFERENCES:
- [Derived] Tomic TJ, Savic AM, Vidakovic AS, Rodic SZ, Isakovic MS, Rodriguez-de-Pablo C, Keller T, Konstantinovic LM. ArmAssist Robotic System versus Matched Conventional Therapy for Poststroke Upper Limb Rehabilitation: A Randomized Clinical Trial. Biomed Res Int. 2017;2017:7659893. doi: 10.1155/2017/7659893. Epub 2017 Jan 31. PMID 28251157